CLINICAL TRIAL: NCT04368364
Title: A Randomized Control Trial Comparing Analgesic Benefits of Ultrasound-guided Single vs Continuous Quadratus Lumborum Blocks vs Intrathecal Morphine for Post Cesarean Section Pain
Brief Title: A Randomized Control Trial Comparing Analgesic Benefits of Ultrasound-guided Single vs Continuous Quadratus Lumborum Blocks (QLB)vs Intrathecal Morphine(ITM) for Post Cesarean Section Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped early due to a conflicting study in the same patient population at the study location.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sudipta Sen, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSC-MS-20-0143
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Pain, Postoperative
Keywords: post c section pain; pain control after baby; nerve block for post delivery pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Control group) (Active Comparator)
  Interventions: Drug: Intrathecal morphine sulfate (ITM)
- Group 2(Bupivacaine hydrochloride group) (Experimental)
  Interventions: Drug: Bupivacaine hydrochloride
- Group 3 (ropivacaine hydrochloride group) (Experimental)
  Interventions: Drug: ropivacaine hydrochloride

INTERVENTIONS:
Drug: Intrathecal morphine sulfate (ITM) — Spinal anesthesia with ITM + US guided QLB single shot sham block + QLB catheters with no continuous infusion
  Arms: Group 1 (Control group)
Drug: Bupivacaine hydrochloride — Spinal anesthesia without ITM + US guided QLB single shot with bupivacaine hydrochloride + QLB catheters with no continuous infusion
  Arms: Group 2(Bupivacaine hydrochloride group)
Drug: ropivacaine hydrochloride — Spinal anesthesia without ITM + US guided QLB single shot with bupivacaine hydrochloride + QLB catheters continuously infusing 0.2% ropivacaine hydrochloride
  Arms: Group 3 (ropivacaine hydrochloride group)

SUMMARY:
the purpose of this study is to compare opioid consumption in morphine equivalents between the groups that received postoperative analgesia with intrathecal morphine versus US guided QL blocks versus US guided QL catheters

ELIGIBILITY:
Inclusion Criteria:

* Elective C section via Pfannenstiel incision
* Living singleton pregnancy
* Gestation week at least 37 weeks
* American Society of Anesthesiologists (ASA) status 1, 2 and 3
* Primary and secondary C sections

Exclusion Criteria:

* Chronic pain
* Opioid tolerant patients
* Allergy to drugs used in the study.
* Cognitive dysfunction
* BMI > 40
* Coagulation disorder
* Local infection
* Inability to tolerate oral medication
* Previous intra-abdominal surgery
* Patients who will receive a combined spinal epidural for their C section
* Local anesthetics injected at any other fascial plane except the QLB plane (for e.g.- local wound infiltration by surgeon)
* Patients who received sedation or general anesthesia during their C section (midazolam, ketamine, fentanyl, propofol, hydromorphone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudipta Sen, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Memorial Hermann Hospital TMC, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Started | 1 | 1 | 1
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group) | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (0) | 33 (0) | 36 (0) | 31.66 (5.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Narcotic Consumption in Morphine Equivalents (in Milligrams)
Description: Total narcotic consumption in morphine equivalents (in milligrams) for the first 72 hours after surgery was calculated.
Time Frame: upto 72 hours post surgery
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
milligrams | 25 (0) | 12.5 (0) | 0 (0)

2. Secondary Outcome: Total Narcotic Consumption in Morphine Equivalents (in Milligrams)
Description: Total narcotic consumption in morphine equivalents (in milligrams) for 12, 24 and 48 hours after surgery was calculated.
Time Frame: 12,24,48 hours post surgery
Population: Data were not collected at 12 hours post surgery.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
milligrams
  12 hours: number analyzed (Participants) | 0 | 0 | 0
  24 hours | 12.5 (0) | 12.5 (0) | 0 (0)
  48 hours | 25 (0) | 12.5 (0) | 0 (0)

3. Secondary Outcome: Static Pain as Measured by the Numerical Pain Score (NPS)
Description: To assess static pain scores, NPS will be recorded while the participant is supine in bed. NPS is a 11-point scale with a higher number indicating more severe pain (total score ranges from 0 to 10).
Time Frame: 6, 12, 24, 48 and 72 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  6 hours | 0 (0) | 2 (0) | 1 (0)
  12 hours | 0 (0) | 4 (0) | 0 (0)
  24 hours | 3.5 (0) | 4 (0) | 2 (0)
  48 hours | 2 (0) | 2 (0) | 2 (0)
  72 hours | 4 (0) | 1 (0) | 1 (0)

4. Secondary Outcome: Severity of Pruritus as Assessed by a Scale
Description: This numeric scale is a 11-point scale with a higher number indicating an extremely severe side effect. Total score ranges from 0 to 10.
Time Frame: 24, 48 and 72 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  24 hours | 6 (0) | 2 (0) | 0 (0)
  48 hours | 0 (0) | 1 (0) | 0 (0)
  72 hours | 0 (0) | 0 (0) | 0 (0)

5. Secondary Outcome: Severity of Nausea as Assessed by a Scale
Description: as for outcome 4
Time Frame: 24, 48 and 72 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  24 hours | 0 (0) | 2 (0) | 0 (0)
  48 houts | 0 (0) | 0 (0) | 0 (0)
  72 hours | 0 (0) | 0 (0) | 0 (0)

6. Secondary Outcome: Severity of Vomiting as Assessed by a Scale
Description: as for outcome 4
Time Frame: 24, 48 and 72 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  24 hours | 0 (0) | 3 (0) | 0 (0)
  48 hours | 0 (0) | 0 (0) | 0 (0)
  72 hours | 0 (0) | 0 (0) | 0 (0)

7. Secondary Outcome: Severity of Sedation as Assessed by a Scale
Description: as for outcome 4
Time Frame: 24, 48 and 72 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  24 hours | 0 (0) | 3 (0) | 0 (0)
  48 hours | 0 (0) | 1 (0) | 1 (0)
  72 hours | 0 (0) | 0 (0) | 0 (0)

8. Secondary Outcome: Patient Satisfaction as Assessed by Likert Scale
Description: Patient reported a score for each of 4 different aspects of satisfaction: their quality of sleep, ability to ambulate, ability to breast or formula feed, and ability to feed and take care of newborn.
  Each of the 4 aspects of satisfaction were rated on a 5-point Likert scale as follows: Extremely satisfied (5), Very satisfied (4), Moderately satisfied (3), Slightly satisfied (2), Not satisfied (1).
Time Frame: 24 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  quality of sleep | 4 (0) | 3 (0) | 4 (0)
  ability to ambulate | 2 (0) | 3 (0) | 5 (0)
  ability to breast or formula feed | 4 (0) | 3 (0) | 5 (0)
  ability to feed and take care of newborn at 24 hours | 3 (0) | 3 (0) | 5 (0)

9. Secondary Outcome: Dynamic Pain as Measured by the Numerical Pain Score (NPS)
Description: To assess dynamic pain scores, the participant be asked to sit up in bed from supine to sitting, and the NPS will then be recorded. If the participant is ambulating, the dynamic pain score during ambulation (rather during sitting) will be assessed. NPS is a 11-point scale with a higher number indicating more severe pain (total score ranges from 0 to 10).
Time Frame: 6, 12, 24, 48 and 72 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  6 hours | 0 (0) | 3 (0) | 1 (0)
  12 hours | 6 (0) | 6 (0) | 1 (0)
  24 hours | 8 (0) | 6 (0) | 2 (0)
  48 hours | 4 (0) | 2 (0) | 2 (0)
  72 hours | 7 (0) | 1 (0) | 1 (0)

10. Secondary Outcome: Patient Satisfaction as Assessed by Likert Scale
Description: as for outcome 8
Time Frame: 48 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  quality of sleep | 4 (0) | 4 (0) | 5 (0)
  ability to ambulate | 4 (0) | 4 (0) | 5 (0)
  ability to breast or formula feed | 4 (0) | 3 (0) | 5 (0)
  ability to feed and take care of newborn at 24 hours | 4 (0) | 4 (0) | 4 (0)

11. Secondary Outcome: Patient Satisfaction as Assessed by Likert Scale
Description: as for outcome 8
Time Frame: 72 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  quality of sleep | 3 (0) | 5 (0) | 5 (0)
  ability to ambulate | 2 (0) | 4 (0) | 5 (0)
  ability to breast or formula feed | 3 (0) | 4 (0) | 5 (0)
  ability to feed and take care of newborn | 3 (0) | 4 (0) | 5 (0)

12. Secondary Outcome: Time to First Analgesic Request
Time Frame: 72 hours post surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
Number analyzed (Participants) | 1 | 1 | 1
minutes | 414 (0) | 1043 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Group 1 (Control Group) | Group 2(Bupivacaine Hydrochloride Group) | Group 3 (Ropivacaine Hydrochloride Group)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Control Group) (N=1) | Group 2(Bupivacaine Hydrochloride Group) (N=1) | Group 3 (Ropivacaine Hydrochloride Group) (N=1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nausea (General disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Sedation (General disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT04368364/Prot_SAP_000.pdf